CLINICAL TRIAL: NCT06856005
Title: "Assessing the Impact of Personalized Music Playlists on Procedural Anxiety and Crown Preparation Performance Among Young Dentists: A Randomized Controlled Trial"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Maria Shakoor Abbasi, Associate Professor, Pakistan Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SOD/ERB/2025/61
Record Dates: First submitted 2025-02-12; First posted 2025-03-04 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Crown; Procedural Anxiety

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): which listened to personalized music during the procedure
  Interventions: Other: Music intervention
- Group B (No Intervention)

INTERVENTIONS:
Other: Music intervention — to evaluate the effectiveness of personalized music playlists in reducing procedural anxiety among young dentists performing crown preparations for porcelain-fused-to-metal (PFM) crowns and to compare the crown preparation performance of students who listened to music with those who did not.
  • Experimental Group:
  o Participants in the experimental group were asked to use personalized music playlists during the procedure. These playlists were already available on their personal devices (e.g., smartphones) and reflected their individual music preferences. Participants selected music they found relaxing or enjoyable, ensuring the intervention was tailored to their unique tastes.
  Arms: Group A

SUMMARY:
The objective of this study was to evaluate the effectiveness of personalized music playlists in reducing procedural anxiety among young dentists performing crown preparations for porcelain-fused-to-metal (PFM) crowns.

A randomized controlled trial with a parallel-group design was conducted at the Department of Prosthodontics, School of Dentistry, Shaheed Zulfiqar Ali Bhutto Medical University, from April 12th, 2024, to October 11th, 2024. A total of 64 young dentists (20-30 years old) were randomly assigned to two groups: the experimental group (Group A), which listened to personalized music during the procedure, and the control group (Group B), which received no music. Anxiety was measured using the State-Trait Anxiety Inventory (STAI) before and after the procedure. Physiological parameters, including heart rate and respiratory rate, were also monitored. The preparation was evaluated based on a structured scoring rubric, assessing critical parameters. The scoring was conducted by two experienced prosthodontists who were blinded to the participant's group allocation. Statistical analysis was performed using SPSS version 25.0.0, with a p-value of <0.05 considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female
* Young dentists 20-30 years.
* Recently graduated from dental school. (graduated within the last 1-3 years.)
* No hearing impairments or known psychiatric disorders.

Exclusion Criteria:

* Dentists with previous experience in anxiety management techniques.
* Those who have already participated in similar studies.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2024-04-12 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Anxiety Assessment: trait and state anxiety. | 2 minutes after the procedure
  The State-Trait Anxiety Inventory (STAI) was used to measure it
Crown preparation was evaluated based on a structured scoring rubric, assessing critical parameters | 2 minutes after the procedure
  The preparation was evaluated based on a structured scoring rubric, assessing critical parameters. The scoring was conducted by two experienced prosthodontists who were blinded to the participant's group allocation

SECONDARY OUTCOMES:
Heart rate was recorded before and after the procedure. | immediately after the procedure
  Heart rate was recorded before and after the procedure.
Respiratory rate was recorded before and after the procedure. | immediately after the procedure
  respiratory rate was recorded before and after the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- School of dentistry, SZABMU, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided